CLINICAL TRIAL: NCT03411785
Title: Evaluation of the Comprehensive Primary Care Plus (CPC+) Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CPCPlus2017
Record Dates: First submitted 2017-09-05; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: All Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPC+ practices (Experimental): This is the intervention group, and includes the practices that were selected and agreed to participate in the CPC+ model.
  Interventions: Other: CPC+ model
- Comparison practices (No Intervention): Comparison practices are the control group. This group includes practices not participating in the model that were matched to the CPC+ practices and whose outcomes will be compared to those of the CPC+ practices.

INTERVENTIONS:
Other: CPC+ model — CPC+ practices receive a monthly care management fee and prospective performance-based incentive payment on top of traditional payments. Some practices will also receive some payment that shifts away from fee-for-service. In addition, CPC+ practices will receive learning and health IT support and data feedback to implement processes to meet care delivery requirements and achieve five primary care functions.
  Arms: CPC+ practices

SUMMARY:
The Comprehensive Primary Care Plus (CPC+) Model, sponsored by the Centers for Medicare & Medicaid Services (CMS), is a multipayer advanced primary care model. CPC+ aims to strengthen primary care by transforming how primary care practices deliver care, supported by regionally based multipayer payment reform, learning support, data feedback, and health information technology (health IT) support. The CPC+ evaluation will assess how CPC+ was implemented; how practices transformed care; and the effects on cost, service use, quality of care, and the experiences of patients, primary care practitioners, and staff. The evaluation will also identify facilitators and barriers to implementation and improved outcomes.

DETAILED DESCRIPTION:
This project is a large, seven-year mixed-methods evaluation of the Comprehensive Primary Care Plus (CPC+) Model, sponsored by the Centers for Medicare & Medicaid Services (CMS). CPC+ aims to improve the delivery of primary care; patients' cost, service use, and quality of care; and the experiences of patients, practitioners, and staff. It aims to achieve these goals by helping practices transform across five key care delivery functions: (1) access and continuity, (2) care management, (3) comprehensiveness and coordination, (4) patient and caregiver engagement, and (5) planned care and population health.

The national model includes two rounds, each of which will last for five years. Round 1 will take place from January 2017 through December 2021 and Round 2 from January 2018 through December 2022. A total of 2,877 primary care practices are participating in Round 1. The number of Round 2 practices will not be confirmed until September 2017.

From practices that applied to participate, CMS selected those that provide primary care, met specific certified health information technology (health IT) requirements, and were already engaging in certain care delivery activities. The CPC+ model includes two transformation tracks with incrementally advanced care delivery requirements and payment options. Participating practices will receive financial payments from CMS, including a monthly care management fee and prospective performance-based incentive payment, on top of traditional payments. Some practices will also receive some payment that shifts away from fee-for-service. In addition, practices will receive payments from other participating payers, representing a large proportion of their total revenue. CPC+ practices will receive learning support, data feedback, and health IT support to promote transformation.

To estimate the effect of CPC+, the investigators will compare the outcomes over time for CPC+ practices with the outcomes over time for a group of comparison practices. The investigators selected the comparison practices by identifying practices that matched the CPC+ practices on key characteristics. The investigators expect to include up to 8,397 comparison practices in Round 1.

The investigators will estimate the impact of CPC+ on patient outcomes by tracking the patients who are attributed to a study practice based on receiving most of their evaluation and management care from that practice. The investigators expect to include approximately 5,326,531 attributed patients across the CPC+ and comparison practices in Round 1 (the number of attributed patients for the Round 2 practices is to be determined). Analyses of Medicare (and in some regions Medicaid) claims data for patients attributed to the CPC+ and comparison practices will be conducted to estimate impacts on Medicare expenditures, our primary outcome, and service use and quality of care.

The investigators will also estimate the impact of CPC+ on practice care delivery approaches, and patient, practitioner, and staff experience. The investigators will administer a practice survey to the practice managers of all the study practices to track changes in care delivery and practice characteristics. The investigators will measure patient experience through a survey administered to Medicare fee-for-service beneficiaries attributed to the study practices. Changes in work environment and practitioner and staff experience with CPC+ will be measured through a survey of primary care practitioners of the study practices and staff of the CPC+ practices. For the Round 1 practices, the investigators expect to administer 11,244 practice surveys, 20,000 patient surveys, 10,996 practitioner surveys, and 10,429 staff surveys, The sample sizes for surveys for the Round 2 practices are to be determined. Telephone interviews and site visits will be conducted with CPC+ payers; practitioners and staff in the practices, and, if relevant, the systems and medical groups that own them; patients; and other stakeholders to understand what was implemented, and barriers and facilitators to implementation and improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All Medicare fee-for-service patients who receive the largest share of their evaluation and management visits from one of the study primary care practices.
* Practice managers, practitioners, and staff of the study primary care practices.

Exclusion Criteria: None

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5326531 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Total Part A and Part B claims paid by Medicare in 2017 | 12 months
  Total claims paid by Medicare for for physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Total Part A and Part B claims paid by Medicare in 2018 | 24 months
  Total claims paid by Medicare for physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Total Part A and Part B claims paid by Medicare in 2019 | 36 months
  Total claims paid by Medicare for physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Total Part A and Part B claims paid by Medicare in 2020 | 48 months
  Total claims paid by Medicare for physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Total Part A and Part B claims paid by Medicare in 2021 | 60 months
  Total claims paid by Medicare for physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health

SECONDARY OUTCOMES:
Claims paid by Medicare in 2017 by type of service and service utilization | 12 months
  Claims paid by Medicare for each of following: physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Claims paid by Medicare in 2018 by type of service and service utilization | 24 months
  Claims paid by Medicare for each of following: physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Claims paid by Medicare in 2019 by type of service and service utilization | 36 months
  Claims paid by Medicare for each of following: physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Claims paid by Medicare in 2020 by type of service and service utilization | 48 months
  Claims paid by Medicare for each of following: physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Claims paid by Medicare in 2021 by type of service and service utilization | 60 months
  Claims paid by Medicare for each of following: physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Claims paid by Medicaid in 2017 | 12 months
  Claims paid by Medicaid for physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Claims paid by Medicaid in 2018 | 24 months
  Claims paid by Medicaid for physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Claims paid by Medicaid in 2019 | 36 months
  Claims paid by Medicaid for physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Claims paid by Medicaid in 2020 | 48 months
  Claims paid by Medicaid for physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Claims paid by Medicaid in 2021 | 60 months
  Claims paid by Medicaid for physician services (primary care physician services, specialist services, and services provided by noninstitutional providers), inpatient hospital services, outpatient services, skilled nursing facility, durable medical equipment, hospice, and home health
Quality-of-care process measures for 2017 based on claims data | 12 months
  Quality-of-care outcome measures based on claims data (including 30-day hospital readmissions, rate of hospitalizations for ambulatory care sensitive admissions, and likelihood of emergency department revisits)
Quality-of-care process measures for 2018 based on claims data | 24 months
  Quality-of-care outcome measures based on claims data (including 30-day hospital readmissions, rate of hospitalizations for ambulatory care sensitive admissions, and likelihood of emergency department revisits)
Quality-of-care process measures for 2019 based on claims data | 36 months
  Quality-of-care outcome measures based on claims data (including 30-day hospital readmissions, rate of hospitalizations for ambulatory care sensitive admissions, and likelihood of emergency department revisits)
Quality-of-care process measures for 2020 based on claims data | 48 months
  Quality-of-care outcome measures based on claims data (including 30-day hospital readmissions, rate of hospitalizations for ambulatory care sensitive admissions, and likelihood of emergency department revisits)
Quality-of-care process measures for 2021 based on claims data | 60 months
  Quality-of-care outcome measures based on claims data (including 30-day hospital readmissions, rate of hospitalizations for ambulatory care sensitive admissions, and likelihood of emergency department revisits)
Patient experience | 24 months
  Self-reported measures of patient experience with primary care practitioner and practice
Patient experience | 36 months
  Self-reported measures of patient experience with primary care practitioner and practice
Patient experience | 60 months
  Self-reported measures of patient experience with primary care practitioner and practice
Practitioner and staff experience | 24 months
  Self-reported measures of approaches to delivery of primary care and work experience at practice
Practitioner and staff experience | 48 months
  Self-reported measures of approaches to delivery of primary care and work experience at practice
Practice's care delivery | 12 months
  Self-reported measures of practice approaches to delivery of primary care
Practice's care delivery | 24 months
  Self-reported measures of practice approaches to delivery of primary care
Practice's care delivery | 36 months
  Self-reported measures of practice approaches to delivery of primary care
Practice's care delivery | 48 months
  Self-reported measures of practice approaches to delivery of primary care
Practice's care delivery | 60 months
  Self-reported measures of practice approaches to delivery of primary care

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Peikes, Ph.D., Study Director — Mathematica Policy Research

IPD SHARING:
Plan to Share IPD: No